CLINICAL TRIAL: NCT04449328
Title: Induced Motion Illusions Through Vision and Tendon Vibrations: Study of Interactions in Hemiplegic Subjects
Acronym: OPTIVIBE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of inclusion
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19CH113; 2019-A01673-54 (Other: ANSM)
Record Dates: First submitted 2020-06-22; First posted 2020-06-26 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Hemiplegia
Keywords: Computerized Mirror Therapy (CMT); Intensive Visual Simulation3 (IVS3); Vibration; Vibrasens; Upper limb rehabilitation; Stroke; Hemiplegic
MeSH Terms: conditions — Hemiplegia; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with first stroke causing hemiplegic (Experimental): Patient with first stroke causing hemiplegic will be included.
  They will have Computerized Mirror Therapy (CMT) associated at tendon vibration:
  * Visit 1: wrist flexion (right and left arms) with 5 randomized experimental conditions (vision+vibration, vision alone, vibration alone, static image+vibration, vision of extension+vibration(incongruence))
  * Visit 2 (1 week later): wrist extension (right and left arms) with 5 randomized experimental conditions (vision+vibration, vision alone, vibration alone, static image+vibration, vision of flexion+vibration (incongruence)) These conditions will be recording by the Kinovea software, which allows the measurement of angles and amplitudes.
  Interventions: Device: Computerized Mirror Therapy (CMT); Device: Tendon vibration
- healthy subjects (Sham Comparator): Healthy subjects will be included.
  They will have Computerized Mirror Therapy (CMT) associated at tendon vibration:
  * Visit 1: wrist flexion (right and left arms) with 5 randomized experimental conditions (vision+vibration, vision alone, vibration alone, static image+vibration, vision of extension+vibration(incongruence))
  * Visit 2 (1 week later): wrist extension (right and left arms) with 5 randomized experimental conditions (vision+vibration, vision alone, vibration alone, static image+vibration, vision of flexion+vibration (incongruence)) These conditions will be recording by the Kinovea software, which allows the measurement of angles and amplitudes.
  Interventions: Device: Computerized Mirror Therapy (CMT); Device: Tendon vibration

INTERVENTIONS:
Device: Computerized Mirror Therapy (CMT) — Computerized Mirror Therapy (CMT) will be realizing by the device Intensive Visual Simulation 3 (IVS3).
  The patient looks on a screen in front of him, mirroring the movements made by his hand, while attempting to perform the same movement with his other hand.
  Other Names: Intensive Visual Simulation3 (IVS3), Dessintey, Saint Etienne, France
Device: Tendon vibration — Transcutaneous vibrations are used. This device allows vibrations from 50 to 120 Hz with amplitude of 1 mm. This study the frequency used is 70 and 80 Hz.
  Other Names: Vibrasens, VB115, Techno Concept, France

SUMMARY:
Two movement illusion techniques can currently be used in clinical practice for motor rehabilitation after stroke hemiplegia: visual illusion (mirror therapy) and proprioceptive illusion (tendon vibration). Mirror therapy, in its computerized version (IVS3, Dessintey, Saint-Etienne, France), is based on the substitution of the deficient visual feedback by a visual feedback of a correctly realized movement. The proprioceptive illusion is based on the external application of a vibrator on muscle tendons at a frequency between 50 and 120 Hz. These two techniques are currently used independently. They are, in theory, complementary and additive. No study has described the combinatorial properties of the illusions generated by these 2 techniques in hemiplegic subjects and healthy subjects.

DETAILED DESCRIPTION:
The study hypothesis is that the administration of mirror therapy together with vibration will increase the perception of movement in a subjective scale.

ELIGIBILITY:
Inclusion Criteria:

Hemiplegic subjects :

* Male or female
* Aged 18 to 70 years,
* First ischemic or hemorrhagic stroke causing hemiplegic
* Having signed the written consent
* Affiliated or entitled to a social security scheme

Healthy subjects :

* Male or female, aged 18 to 70 years,
* Matched in sex, age and laterally with hemiplegic subjects
* Having signed the written consent
* Affiliated or entitled to a social security scheme

Exclusion Criteria:

Hemiplegic subjects :

* With complete lesion of the primary motor cortex
* With an addiction to alcohol or drugs
* With psychiatric illness, cognitive impairment, uncontrolled disease/epilepsy, malignant illness severe kidney or lung disease
* With history of associated general disabling disease
* With cerebellar syndrome
* With clinical brain stem involvement
* Under legal protection
* Pregnant or breastfeeding women

Healthy subjects :

* Neurological, cardiovascular, musculoskeletal diseases
* Taking medication that can affect attention
* Unable to understand instructions of the study
* Under legal protection
* Pregnant or breastfeeding women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
subjective measure of the intensity of the perception of movements: change from baseline impression of movement at day 7 | Day: 0, 7
  Measured impression of movement on conditions (visual and/or proprioceptive; yes/no/don't know)
subjective measure of the intensity of the perception of movements: change from baseline nature of this impression at day 7 | Day: 0, 7
  Measured nature of this impression of movement (flexion/extension)
subjective measure of the intensity of the perception of movements: change from baseline intensity of the movement felt at day 7 | Day: 0, 7
  Measured intensity of the movement felt by Visual Analogue Scale (VAS) results (0 = no sense of movement and 10 = like real movement.)

SECONDARY OUTCOMES:
Objective measurement of the perceived movement angle reproduced without motor intention by the hemiplegic subjects with the healthy limb | Day: 0, 7
  Measured by Kinovea software.
Measurement of motor intention in hemiplegic subjects by experimental conditions | Day: 0, 7
  Measured by Visual Analogue Scale (VAS) results (0 = no sense of movement and 10 = like real movement).
To compare the Visual Analogue Scale (VAS) score according to the level of motor impairment | Day: 0
  Level of motor impairment is measured by Medical Research Council (MRC) score. Medical Research Council (MRC) score evaluate motricity (0= paralyzed).
To compare the Visual Analogue Scale (VAS) score with the Erasmus modified Nottingham Sensory Assessment (EmNSA) score | Day: 0
  Erasmus modified Nottingham Sensory Assessment (EmNSA) score evaluated the level of sensory impairment.
  The Erasmus modified Nottingham Sensory Assessment (EmNSA) includes 2 subscales: somatosensory score (min 0 and max 44) and stereognosis (min 0 and max 20) for left and right members.
Intensity of the perception of movements using a visual analogue scale and the objective measurement of perceived movement angle reproduced by the healthy subjects with the vibrated arm | Day: 0, 7
  Measured by Kinovea software.
Brain activity according to different experimental conditions (with and without vibration or with and without visual illusion) in hemiplegic subjects. | Day: 0, 7
  Multi Channel EEG Acquisition System

CONTACTS AND LOCATIONS:
Overall Officials: Pascal GIRAUX, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adham A, Bessaguet H, Struber L, Rimaud D, Ojardias E, Giraux P. Distinct and additive effects of visual and vibratory feedback for motor rehabilitation: an EEG study in healthy subjects. J Neuroeng Rehabil. 2024 Sep 12;21(1):158. doi: 10.1186/s12984-024-01453-3. PMID 39267092